CLINICAL TRIAL: NCT00023075
Title: Nuclear Magnetic Spectroscopy for the Evaluation of Primary Lateral Sclerosis, Hereditary Spastic Paraplegia and Amyotrophic Lateral Sclerosis
Brief Title: Nuclear Magnetic Spectroscopy Imaging to Evaluate Primary Lateral Sclerosis, Hereditary Spastic Paraplegia and Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010241; 01-N-0241
Record Dates: First submitted 2001-08-22; First posted 2001-08-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-08

CONDITIONS: Primary Lateral Sclerosis; Hereditary Spastic Paraplegia; Amyotrophic Lateral Sclerosis
Keywords: MRI; Neuromuscular Disease; N-Acetyl Aspartate; Choline; Creatine; Spasms; Spasticity; Primary Lateral Sclerosis; Hereditary Spastic Paraplegia; Spastic Paraparesis; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Motor Neuron Disease; Spastic Paraplegia, Hereditary; Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Spasm; Muscle Spasticity; Paraparesis, Spastic

SUMMARY:
This study will use a magnetic resonance imaging technique called nuclear magnetic spectroscopy (H-MRS) to define the pathology and progression of primary lateral sclerosis, hereditary spastic paraplegia and amyotrophic lateral sclerosis and assess the usefulness of this technique in evaluating patients' response to therapy. H-MRS will be used to examine metabolic changes in the parts of the brain and spinal cord (motor cortex and corticospinal tract) involved in movement.

Normal volunteers and patients with primary lateral sclerosis, hereditary spastic paraplegia or amyotrophic lateral sclerosis between 21 and 65 years of age may be eligible for this study. Participants will have up to five H-MRS studies, including baseline and follow-up tests. For this procedure, the subject lies on a stretcher that is moved into a strong magnetic field. Earplugs are worn to muffle the loud knocking noise that occurs during switching of radio frequencies. The subject will be asked to lie still during each scan, for 1 to 8 minutes at a time. Total scanning time varies from 20 minutes to 2 hours, with most examinations lasting between 45 and 90 minutes. Communication with the medical staff is possible at all times during the scan.

DETAILED DESCRIPTION:
Standard MRI imaging of the brain shows no consistent abnormalities in many degenerative disorders with progressive upper motor neuron symptoms, including primary lateral sclerosis, hereditary spastic paraparesis, and amyotrophic lateral sclerosis. Nuclear magnetic resonance spectroscopy (H-MRS) is able to evaluate certain cerebral metabolites that reflect the functioning and integrity of neurons. The objective of this protocol is to study metabolic changes in the motor cortex and corticospinal tract using MRS in these disorders to characterize the pathology, the progression of the diseases, and assess the utility of MRS to follow the response to therapies.

ELIGIBILITY:
INCLUSION CRITERIA:

Adult patients with PLS, HSP, and ALS already evaluated by protocol #01-N-0148.

Adult normal volunteers

EXCLUSION CRITERIA:

Pregnancy, implanted devices such as pacemakers, medication pumps or defibrillators, metal in the cranium except the mouth, intracardiac lines, history of eye shrapnel injury or any other condition/device that may contraindicate or prevent the acquisition of an MRI.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55
Dates: Start 2001-08; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bonneau D, Rozet JM, Bulteau C, Berthier M, Mettey R, Gil R, Munnich A, Le Merrer M. X linked spastic paraplegia (SPG2): clinical heterogeneity at a single gene locus. J Med Genet. 1993 May;30(5):381-4. doi: 10.1136/jmg.30.5.381. PMID 8320699
- [Background] Chan S, Shungu DC, Douglas-Akinwande A, Lange DJ, Rowland LP. Motor neuron diseases: comparison of single-voxel proton MR spectroscopy of the motor cortex with MR imaging of the brain. Radiology. 1999 Sep;212(3):763-9. doi: 10.1148/radiology.212.3.r99au35763. PMID 10478245
- [Background] Comi G, Rovaris M, Leocani L. Review neuroimaging in amyotrophic lateral sclerosis. Eur J Neurol. 1999 Nov;6(6):629-37. doi: 10.1046/j.1468-1331.1999.660629.x. PMID 10529749